CLINICAL TRIAL: NCT06228833
Title: A Prospective, Single-center, Single-blind, Randomized Split-face Controlled Clinical Study to Evaluate the Efficacy and Safety of Monopolar Radiofrequency Combined With SkinCeuticals A.G.E and Skinceuticals CE FERULIC for Improving Facial Skin Elasticity, Tightening and Fading Fine Lines
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of Monopolar Radiofrequency Combined With SkinCeuticals A.G.E and Skinceuticals CE FERULIC for Improving Facial Skin Elasticity, Tightening and Fading Fine Lines
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yes Skin Medical Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SKCRFAGE002
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Skin Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental)
  Interventions: Device: monopolar radiofrequency; Other: SkinCeuticals A.G.E and Skinceuticals CE FERULIC
- Control group (Active Comparator)
  Interventions: Device: monopolar radiofrequency; Other: Standard Cream

INTERVENTIONS:
Device: monopolar radiofrequency — Each subject underwent monopolar radiofrequency treatment (Thermage FLX ™ ) on both sides of the face
Other: SkinCeuticals A.G.E and Skinceuticals CE FERULIC — Test Side receives SkinCeuticals A.G.E and Skinceuticals CE FERULIC
  Arms: Test group
Other: Standard Cream — Control Side applies Standard Cream
  Arms: Control group

SUMMARY:
A Prospective, Single-center, Single-blind, Randomized split-face, controlled trial will be conducted. The goal of this clinical trial is to evaluate the efficacy and safety of monopolar radiofrequency combined with SkinCeuticals A.G.E and Skinceuticals CE FERULIC for improving facial skin elasticity, tightening and fading fine lines

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to be enrolled in the study:

  1. Healthy women, skin quality is not limited, aged 25 ~ 65 years old face old ~ moderate aging group;
  2. subjects facial skin rough, loose, lack of elasticity;
  3. Subjects with multiple facial fine lines, decree lines or puppet lines areas have static fine lines trend, the lower part showed signs of loosening;
  4. Subjects with consistent facial skin status on both sides and planning to receive monopolar radiofrequency treatment;
  5. Be able to cooperate well with the tester and maintain the regularity of life during the study;
  6. Be able to read and understand all contents of the informed consent form, and voluntarily sign the informed consent form (ICF);
  7. Agreed not to use any cosmetics, drugs and health products that have an impact on the results during the trial;

Exclusion Criteria:

* Subjects were not included in the study if they met any of the following exclusion criteria:

  1. Subjects with contraindications to monopolar radiofrequency treatment (such as malignant tumors, acute systemic infection, metal implants or active implants in the body such as cardiac pacemakers/defibrillators, etc.) or contraindications to A.G.E./CE use (or allergies to other skin care components);
  2. Subjects with facial skin diseases, infections, inflammation, etc. that may affect the judgment of the test results;
  3. Subjects with hypertrophic scar or scar constitution;
  4. Subjects who have experienced tightening medical treatment (Gemma, Fotona 4D, ultrasonic cannon, ultrasonic scalpel, gold microneedle, etc.) in the past 3 months;
  5. Subjects who have oral and topical cosmetic products that may affect the study results within 2 weeks;
  6. Subjects who participate in drug clinical trials or other trials within 30 days, or subjects who have systemic use of drugs that may affect the study results within the past 1 week;
  7. Pregnant or lactating women, or recent plans to prepare for pregnancy;
  8. Other subjects who are not suitable for participating in this study as assessed by the investigator.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Global aesthetic improvement scale （GAIS） score | at day 90 after procedure
  Investigator Satisfaction Assessment Form. Scoring criteria: 3 (very much improved), 2 (marked improvement), 1 (improved), 0 (no change), or -1 (worse).

SECONDARY OUTCOMES:
Global aesthetic improvement scale （GAIS） score | at 30, 60 days after procedure
  Investigator Satisfaction Assessment Form. Scoring criteria: 3 (very much improved), 2 (marked improvement), 1 (improved), 0 (no change), or -1 (worse).
Improvement of skin glossiness | at 30, 60, 90 days after procedure
  Skin glossiness was assessed by an independent investigator on both sides of the face (three measurements averaged) according to DermaLab ® Combo (Multipurpose Skin Detector, Cortex) + Chromaticity Test Probe
Improvement in skin elasticity and tightness | at 30, 60, 90 days after procedure
  Skin elasticity was assessed by an independent investigator on both sides of the face (averaged over three measurements) according to the DermaLab ® Combo + Elastic Probe
Improvement in dermal thickness/density | at 30, 60, 90 days after procedure
  Dermal thickness/density was assessed on both sides of the face (averaged over three measurements) by an independent investigator using the DermaLab ® Combo + HF ultrasound probe
Improvement of transepidermal water loss (TEWL) | at 30, 60, 90 days after procedure
  TEWL was assessed by an independent investigator on both sides of the face (three measurements averaged) according to the DermaLab ® Combo + TEWL test probe
Improvement of skin stratum corneum water content | at 30, 60, 90 days after procedure
  Skin stratum corneum moisture was assessed on both sides of the face (three measurements averaged) by an independent investigator using the DermaLab ® Combo + Moisture Testing Probe
Improvement in fine lines score | at 30, 60, 90 days after procedure
  Skin Parameter Assessment Form. Fine lines: Grading was performed on a Griffith 's scale (10-point scale) with different scores representing: 0 (no fine lines/wrinkles, skin completely smooth and no wrinkles); 1-3 (mild, few fine lines and wrinkles, and distant intervals within the treatment area); 4-6 (moderate, moderate number of fine lines/wrinkles within the treatment area and close to each other); and 7-9 (severe, dense clusters of fine lines/wrinkles within the treatment area). Fine lines status should be evaluated by an independent investigator.
Subject satisfaction evaluation | at 30, 60, 90 days after procedure
  Subject Satisfaction Assessment Form. 1: very dissatisfied, 2: dissatisfied, 3: fair, 4: satisfied, and 5: very satisfied, and the proportion of people in each rating was statistically summarized